CLINICAL TRIAL: NCT03640312
Title: A Double Blind Randomized Controlled Trial to Assess the Efficacy and Safety of a Quadruple Ultra-low-dose Treatment for Hypertension (QUARTET USA)
Brief Title: Efficacy and Safety of a Quadruple Ultra-low-dose Treatment for Hypertension
Acronym: QUARTET USA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: ACCESS Community Health Network (Other); University of Sydney (Other)
Responsible Party: Principal Investigator, Mark Huffman, Professor of Medicine and Global Health Center Co-Director, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202203097-STU00205834
Record Dates: First submitted 2018-08-15; First posted 2018-08-21 (Actual); Results first posted 2023-09-22 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Hypertension
Keywords: Hypertension; Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — candesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QUARTET LDQT (Experimental): Patients randomized to the intervention arm will take a once daily ultra-low-dose quadruple combination therapy (QUARTET LDQT). The LDQT is an overencapsulated combination pill comprising four types of blood pressure lowering medications each at ¼ standard doses. QUARTET includes candesartan 2mg, amlodipine besylate 1.25mg, indapamide 0.625mg, and bisoprolol 2.5mg. The individual components are currently approved and marketed within the United States.
  Interventions: Drug: QUARTET LDQT
- Candesartan (Active Comparator): Patients randomized to the comparison arm will take a once daily 8mg candesartan.
  Interventions: Drug: Candesartan

INTERVENTIONS:
Drug: QUARTET LDQT — Ultra-low-dose combination therapy comprising four different blood pressure lowering drugs at 1/4 dosages. Taken once daily for 12 weeks.
  Arms: QUARTET LDQT
Drug: Candesartan — Standard monotherapy of 8mg candesartan. Taken once daily for 12 weeks.
  Arms: Candesartan

SUMMARY:
To investigate, in a double-blind randomized controlled trial, whether initiating treatment with ultra-low-dose quadruple-combination therapy ("LDQT") will lower office blood pressure more effectively, and with fewer side effects, compared to initiating standard dose monotherapy as per current guidelines in patients with hypertension.

Primary hypothesis: A combination pill comprising four types of blood pressure lowering medications, each at one-quarter standard doses, will lower office blood pressure more effectively than initiating patients with standard dose monotherapy as per contemporary clinical practice guideline recommendations.

DETAILED DESCRIPTION:
This trial will investigate whether initiating treatment with ultra-low-dose quadruple-combination therapy (LDQT; including candesartan 2 mg, amlodipine 1.25 mg, indapamide 0.625 mg, and bisoprolol 2.5 mg) will lower automated office blood pressure and 24-hour ambulatory blood pressure at 12 weeks more effectively, and with no increase in side effects, compared to initiating standard dose monotherapy (candesartan 8 mg) in adults with raised blood pressure (SBP>130 mmHg or DBP>80 mmHg) and without cardiovascular disease. Our preliminary data from a short-term (4-week) crossover trial of 18 participants suggest that LDQT lowers office blood pressure by 22/13 mmHg on average compared with placebo with no difference in serious adverse events. Effects on 24-hour ambulatory blood pressure were similar.

The investigators will perform this phase II, single site, randomized controlled trial in a network of federally qualified health centers in Chicago because this population bears a disproportionate burden of blood pressure related diseases, and the investigators have previously successfully conducted clinical studies in this population.

While the investigators hypothesize this intervention will be easily implemented and efficacious for all patients and clinicians, the investigators will explore variation in treatment effect by potential moderating variables, including age, sex, race/ethnicity, and health literacy level. Beyond examining efficacy, the investigators also plan to assess feasibility of implementing this intervention in a clinical setting by simultaneously evaluating implementation outcomes of acceptability, preferences, and lessons of LDQT among patients and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Spanish or English speaker.
* Previous documentation within the past 24 months of hypertension or high blood pressure (SBP 130-179 mmHg or DBP 80-109 mmHg) from general practitioner, pharmacist or health care professional (e.g., medical assistant, physician or nurse).
* Either: 1) Untreated (automated) clinic SBP 140-179 or DBP 90-109 mmHg in the last 12 weeks, OR 2) Monotherapy with clinic SBP 130-159 or DBP 85-99 mmHg in the last 12 weeks.
* Either: 1) Treatment naïve, OR 2) Currently not on treatment (not take in last 4 weeks), OR 3) Currently taking 1 BP lowering drug (ACE, ARB, CCB, thiazide- or thiazide-like diuretic, BB, MRA, alpha blocker) at any dose.
* Research grade blood pressure measurement (baseline mean) SBP>= 115 mmHg and DBP >= 60 mmHg

Exclusion Criteria:

* Known contraindication to candesartan, amlodipine, indapamide or bisoprolol.
* Previous diagnosis of coronary artery disease, stroke, or heart failure.
* Presence of significant proteinuria (based on 3+ proteinuria via spot urinalysis or >300mg/dL of proteinuria based on random urinary albumin-to-creatinine ratio testing of 300 mg/g)
* Evidence of secondary cause of hypertension e.g., renal artery stenosis; significant renal impairment (eGFR <50 ml/min/1.73 m2), raised serum potassium (above lab normal limit of 5.5 mEq/L).
* Women who are pregnant, breast feeding or of childbearing potential and are not using and do not plan to continue using medically acceptable form of contraception throughout the study (pharmacological or barrier methods).
* Concomitant illness, physical impairment or mental condition which in the opinion of the study team / primary care physician could interfere with the conduct of the study including outcome assessments.
* Participation in a concurrent interventional medical investigation or pharmacologic clinical trial. Patients in observational, natural history or epidemiological studies not involving an intervention are eligible.
* Participant's responsible primary care or other responsible physician believes it is not appropriate for participant to switch current monotherapy.
* Inability or unwillingness to provide written informed consent.
* Unable to complete study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Huffman, PhD, MD, Principal Investigator — Northwestern University Feinberg School of Medicine; Jody D Ciolino, PhD, Principal Investigator — Overall Study Officials:
Locations (2):
- United States (2):
  - ACCESS Martin T. Russo Family Health Center, Bloomingdale, Illinois
  - Ashland Family Health Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared through NHLBI BioLINCC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 1 year of study conclusion.
Access Criteria: Access to study data will be managed through NHLBI BioLINCC

REFERENCES:
- [Derived] Huffman MD, Baldridge AS, Lazar D, Abbas H, Mejia J, Flowers FM, Quintana A, Jackson A, Kandula NR, Lloyd-Jones DM, Persell SD, Khan SS, Paparello JJ, Chopra A, Tripathi P, Vu MH, Chow CK, Ciolino JD. Efficacy and safety of a four-drug, quarter-dose treatment for hypertension: the QUARTET USA randomized trial. Hypertens Res. 2024 Jun;47(6):1668-1677. doi: 10.1038/s41440-024-01658-y. Epub 2024 Apr 8. PMID 38584159
- [Derived] Sanuade OA, Jacobson TA, Quintana A, Flowers FM, Abbasi H, Vu MH, Baldridge AS, Mejia J, Lazar D, Ciolino JD, Huffman MD, Kandula NR. Process Evaluation of a Double-Blind Randomized Controlled Trial to Assess the Efficacy and Safety of a Quadruple Ultra-Low-Dose Treatment for Hypertension Within a Federally Qualified Health Center Network (QUARTET USA). J Am Heart Assoc. 2024 Jan 2;13(1):e032236. doi: 10.1161/JAHA.123.032236. Epub 2023 Dec 29. PMID 38156601
- [Derived] Baldridge AS, Huffman MD, Lazar D, Abbas H, Flowers FM, Quintana A, Jackson A, Khan SS, Chopra A, Vu M, Tripathi P, Jacobson T, Sanuade OA, Kandula NR, Persell SD, Paparello JJ, Rosul LL, Mejia J, Lloyd-Jones DM, Chow CK, Ciolino JD. Efficacy and safety of a quadruple ultra-low-dose treatment for hypertension (QUARTET USA): Rationale and design for a randomized controlled trial. Am Heart J. 2022 Dec;254:183-193. doi: 10.1016/j.ahj.2022.09.004. Epub 2022 Sep 15. PMID 36116516

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 120 were consented and assessed for eligibility. 58 were excluded for not meeting either inclusion or exclusion criteria, declining participation, or not showing up for randomization visits. Thus, these 58 individuals were not randomized, and 62 participants were randomized
Pre-assignment Details: NA - all enrolled participants were randomized.
Groups:
- QUARTET LDQT: Patients randomized to the intervention arm took a once daily ultra-low-dose quadruple combination therapy (QUARTET LDQT). The LDQT is an overencapsulated combination pill comprising four types of blood pressure lowering medications each at ¼ standard doses. QUARTET includes candesartan 2mg, amlodipine besylate 1.25mg, indapamide 0.625mg, and bisoprolol 2.5mg. The individual components are currently approved and marketed within the United States.
  QUARTET LDQT: Ultra-low-dose combination therapy comprising four different blood pressure lowering drugs at 1/4 dosages. Taken once daily for 12 weeks.
- Candesartan: Patients randomized to the comparison arm took a once daily 8mg candesartan.
  Candesartan: Standard monotherapy of 8mg candesartan. Taken once daily for 12 weeks.
Period: Overall Study
Arm/Group | QUARTET LDQT | Candesartan
Started | 32 | 30
6 Week Follow Up | 32 | 28
Completed | 29 | 24
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QUARTET LDQT | Candesartan | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (12.6) | 52 (10.5) | 52 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 17 | 17 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 24 | 21 | 45
  Race/Ethnicity: Black/Sub Saharan African | 4 | 7 | 11
  Race/Ethnicity: White/Caucasian/Other | 4 | 2 | 6
Body Mass Index, kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 33 (6.9) | 34 (7.9) | 34 (7.3)
Heart rate, beats per minute [Mean (Standard Deviation); unit: beats per minute] | 71.5 (10.0) | 71.7 (11.7) | 71.6 (10.8)
History of diabetes, n (%) [Count of Participants; unit: Participants] | 10 | 7 | 17
History of smoking, n (%) [Count of Participants; unit: Participants] | 11 | 9 | 20
History of depression, n (%) [Count of Participants; unit: Participants] | 7 | 9 | 16
Weekly alcohol use, n (%) [Count of Participants; unit: Participants] | 10 | 9 | 19
Systolic Blood Pressure, mm Hg [Mean (Standard Deviation); unit: mm Hg] | 137.6 (11.8) | 138.7 (10.8) | 138.1 (11.2)
Diastolic Blood Pressure, mm Hg [Mean (Standard Deviation); unit: mm Hg] | 84.3 (9.6) | 84.3 (11.5) | 84.3 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Systolic Blood Pressure
Description: Mean change (from baseline) in automated office systolic blood pressure adjusted for baseline values.
Time Frame: 12 weeks
Population: Modified intent to treat whereby all those participants with data at any follow-up time point and baseline to contribute to analyses will be included in analyses according to arm to which they were randomized, regardless of adherence to the study protocol.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
mm Hg | -15.65 [-19.70 to -11.60] | -10.87 [-15.24 to -6.50]
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Test type: Superiority; p = 0.114, Mixed Models Analysis — Adjusting for baseline systolic blood pressure; Difference in Least Squared Means (LSM). Random participant effect, fixed baseline, study arm, and time effects; Mean Difference (Net) = -4.78, 95% CI 2-sided [-10.74 to 1.18], Standard Error of Mean 2.97

2. Secondary Outcome: Mean Systolic Blood Pressure
Description: Mean automated office systolic blood pressure adjusted for baseline values.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
mm Hg | 122.37 [118.32 to 126.42] | 127.15 [122.78 to 131.52]
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Test type: Superiority — Adjusted for baseline systolic blood pressure; p = 0.114, Mixed Models Analysis; Mean Difference (Net) = -4.78, 95% CI 2-sided [-10.74 to 1.18], Standard Error of Mean 2.97

3. Secondary Outcome: Change in Mean Diastolic Blood Pressure
Description: Mean change (from baseline) in automated office diastolic blood pressure adjusted for baseline values.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
mm Hg | -11.60 [-14.16 to -9.04] | -6.74 [-9.50 to -3.98]
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Adjusted for baseline diastolic blood pressure; Test type: Superiority; p = 0.012, Mixed Models Analysis — Adjusted Least Squares Mean; Mean Difference (Net) = -4.86, 95% CI 2-sided [-8.62 to -1.11], Standard Error of Mean 1.87

4. Secondary Outcome: Mean Diastolic Blood Pressure
Description: Mean automated office diastolic blood pressure adjusted for baseline values.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
mm Hg | 73.01 [70.46 to 75.57] | 77.88 [75.12 to 80.64]
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Test type: Superiority; p = 0.012, Mixed Models Analysis; Mean Difference (Net) = -4.86, 95% CI 2-sided [-8.62 to -1.11], Standard Error of Mean 1.87

5. Secondary Outcome: Proportion of Patients With Hypertension Control
Description: Proportion of patients with hypertension control (percent with SBP < 130 mmHg and DBP <80 mmHg).
Time Frame: 6 and 12 weeks
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
proportion of participants
  6 weeks | 0.6875 | 0.3929
  12 weeks | 0.6667 | 0.5769
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Test type: Superiority; p = 0.077, Mixed Models Analysis; Generalized Linear Mixed Model (binomial distribution assumption with logit link); Odds Ratio (OR) = 2.40, 95% CI 2-sided [0.91 to 6.35]

6. Secondary Outcome: Number of Patients Requiring Step up Treatment
Description: Number of patients requiring step-up treatment.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
Participants | 6 | 16
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Logistic regression model adjusting for baseline systolic and diastolic blood pressure; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 0.13, 95% CI 2-sided [0.03 to 0.48]

7. Secondary Outcome: Proportion of Patients With Adverse Event Free Hypertension Control
Description: Proportion of patients with adverse event free hypertension control (percent with SBP < 130 mmHg and DBP <80 mmHg).
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 30 | 26
Participants | 6 | 9
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Generalized linear mixed model adjusting for baseline systolic and diastolic blood pressure. Random participant effects. Fixed baseline systolic, diastolic, study arm, and time effects; Test type: Superiority; p = 0.710, Mixed Models Analysis; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.24 to 2.69]

8. Secondary Outcome: Medication Adherence
Description: Medication adherence defined by objective pill counts
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
Participants | 21 | 21
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Logistic regression model adjusting for baseline systolic and diastolic blood pressure; Test type: Superiority; p = 0.437, Regression, Logistic; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.21 to 1.98]

9. Secondary Outcome: Health-related Quality of Life
Description: Mean change (from baseline) in health-related quality of life using Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health instrument. PROMIS Global Health is a gauge of general health-care related quality of life. Possible PROMIS Global Physical Health and Global Mental Health scores range from 0-20, with 20 indicating best possible state of health. Raw scores are converted to T-scores to compare to a standardized population. A PROMIS T-score of 50 represents the mean of the population (SD = 10). Higher values here also indicate better health. A positive change in T score, as reported in this outcome measure, would represent an improvement in Global Physical Health or Global Mental Health at 12 weeks compared to baseline.
Time Frame: 12 weeks
Population: Data are available on only 28 participants in the intervention group for the mental health T score.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 29 | 25
score on a scale
  Change in Physical Health T score (PROMIS) | 1.28 (7.48) | 5.99 (6.97)
  Change in Mental Health T score (PROMIS): number analyzed (Participants) | 28 | 25
  Change in Mental Health T score (PROMIS) | 2.86 (6.25) | 2.76 (7.63)
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Statistical test for difference in Physical Health T Score; Test type: Superiority; p = 0.09, ANCOVA — Adjusted for baseline T score; Mean Difference (Net) = -3.45, 95% CI 2-sided [-7.49 to 0.59], Standard Error of Mean 2.01
Statistical Analysis 2: Comparison: QUARTET LDQT vs Candesartan; Statistical test for difference in Mental Health T Score; Test type: Superiority; p = 0.77, ANCOVA — Adjusted for baseline mental health T score; Mean Difference (Net) = 0.55, 95% CI 2-sided [-3.22 to 4.32], Standard Error of Mean 1.88

10. Secondary Outcome: Change in Mean Systolic Blood Pressure
Description: Mean change (from baseline) in automated office systolic blood pressure adjusted for baseline values.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
mm Hg | -15.65 [-19.70 to -11.60] | -10.87 [-15.24 to -6.50]
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Linear mixed model. Random participant effects. Fixed baseline systolic, study arm, and time effects; Test type: Superiority; p = 0.114, Mixed Models Analysis; Mean Difference (Net) = -4.78, 95% CI 2-sided [-10.74 to 1.182], Standard Error of Mean 2.97

11. Other Pre Specified Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: Percentage of participants with any Serious Adverse Events (SAE) according to Good Clinical Practice definition: adverse events that result in death, are life threatening, require hospitalization or prolong existing hospitalization, result in persistent disability, result in congenital anomaly or birth defect, or unimportant medical event that requires intervention to prevent any of the above.
Time Frame: 12 weeks
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
Participants | 2 | 0
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Test type: Superiority; p = 0.49, Fisher Exact; Risk Difference (RD) = -0.06, 95% CI 2-sided [-0.15 to 0.02], Standard Error of Mean 0.04

12. Other Pre Specified Outcome: Percentage of Participants With Potentially Related Adverse Events
Description: Percentage of participants with occurrence of any potentially related adverse event (pre-specified as in study procedures). Defined as: At least possibly related to study drug.
Time Frame: 12 weeks
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
Participants | 8 | 3
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Test type: Superiority; p = 0.21, Chi-squared; Risk Difference (RD) = -0.15, 95% CI 2-sided [-0.33 to 0.03], Standard Error of Mean 0.09

13. Other Pre Specified Outcome: Rate of Adverse Events of Special Interest
Description: Rate of pre-specified adverse events that are known side effects of active ingredients at the participant level.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
Participants | 16 | 10
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Test type: Superiority; p = 0.18, Chi-squared; Risk Difference (RD) = -0.17, 95% CI 2-sided [-0.41 to 0.08], Standard Error of Mean 0.12

14. Other Pre Specified Outcome: Mean Change in Serum Potassium
Description: Mean change (from baseline) in continuous serum potassium.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
mEq/L | 0.01 (0.42) | 0.02 (0.31)
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Test type: Superiority; p = 0.56, Mixed Models Analysis; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.24 to 0.13], Standard Error of Mean 0.09

15. Other Pre Specified Outcome: Mean Change in Serum Sodium
Description: Mean change (from baseline) in continuous serum sodium.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
mEq/L | -0.81 (2.00) | -0.15 (2.66)
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Test type: Superiority; p = 0.12, Mixed Models Analysis — Linear mixed model. Random participant effects. Fixed baseline systolic, study arm, and time effects; Mean Difference (Net) = -0.71, 95% CI 2-sided [-1.61 to 0.19], Standard Error of Mean 0.45

16. Other Pre Specified Outcome: Mean Change in Blood Urea Nitrogen
Description: Mean change (from baseline) in continuous blood urea nitrogen.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
mg/dL | 0.38 (4.23) | -0.40 (7.11)
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Test type: Superiority; p = 0.94, Mixed Models Analysis — Linear mixed model. Random participant effects. Fixed baseline systolic, study arm, and time effects; Mean Difference (Net) = 0.08, 95% CI 2-sided [-1.84 to 1.99], Standard Error of Mean 0.95 — The model estimated mean differences, adjusted for covariates, will not be equal to the raw mean differences observed

17. Other Pre Specified Outcome: Mean Change in Serum Creatinine
Description: Mean change in continuous serum creatinine.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | QUARTET LDQT | Candesartan
Number analyzed (Participants) | 32 | 30
mg/dL | -0.04 (0.11) | -0.04 (0.11)
Statistical Analysis 1: Comparison: QUARTET LDQT vs Candesartan; Test type: Superiority; p = 0.55, Mixed Models Analysis — Linear mixed model. Random participant effects. Fixed baseline systolic, study arm, and time effects; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.07 to 0.04], Standard Error of Mean 0.03

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Same as clinicaltrials.gov definition.
  A known side effects checklist (included in protocol and consent) was used as a dropdown list for site staff to populate as appropriate at each participant encounter. Any reported side effects from this list were documented as an AE. If an AE did not meet any of these pre-specified terms, the site staff would document 'other' and specify. At specified intervals, a blinded third party MedDRA coder would enter the MedDRA terms into the safety database.
Arm/Group | QUARTET LDQT | Candesartan
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/32 | 0/30
Other Adverse Events (participants affected / at risk) | 20/32 | 14/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QUARTET LDQT (N=32) | Candesartan (N=30)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | NA — Motor Vehicle Accident. Severity: Severe. Outcome: Resolved with sequelae. Blinded relatedness assessment: Unrelated. Investigational product action taken: Temporarily Withdrawn. Resulted in hospitalization.
Chest Pain (General disorders) | 1 (1) | NA — Severity: Severe. Outcome: Resolved with Sequelae. Relatedness Assessment: Unrelated. Investigational Product action taken: Temporarily Withdrawn. Resulted in hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QUARTET LDQT (N=32) | Candesartan (N=30)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) — 2 Total events: 1. Severity: Mild. Outcome: Ongoing at study exit. Relatedness assessment: Unrelated. Investigational product action taken: None. Study arm: Candesartan 2. Severe, resolved without sequelae, unlikely related, no action taken, LDQT
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) — Palpitations, mild, resolved without sequelae, possible relatedness, no IP action taken.
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Ringing in ears, mild, ongoing at study exit, assessed unrelated, no IP action taken.
Eye pruritis (Eye disorders) | 1 (1) | 0 (0) — Itchy eyes, mild, resolved without sequelae, unlikely relatedness, no IP action taken
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) — 5 total events (2 control, 3 LDQT) Diarrhea, mild (5/5), resolved w/o sequelae (4/5) ongoing at study exit (1/5), unlikely (2/5) unrelated (3/5), no IP action taken (4/5) temporarily withdrawn (1/5).
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) — 3 total Stomach cramping (1/3) stomach gas/pain (2/3), mild (3/3), resolved without sequelae (2/3) ongoing at study exit (1/3), unrelated (3/3), no IP action taken (1/3) temporarily withdrawn (1/3) permanently discontinued (1/3)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) — mild, resolved without sequelae, unrelated, no IP action taken
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — mild, resolved without sequelae, unrelated, no IP action taken
Throat irritation (Gastrointestinal disorders) | 1 (1) | 0 (0) — mild, resolved without sequelae, possible relatedness, no IP action taken
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Nausea/vomiting, mild, resolved without sequelae, possible relatedness, permanently discontinued
Dry throat (Gastrointestinal disorders) | 1 (1) | 0 (0) — mild, resolved without sequelae, possible relatedness, temporarily withdrawn
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Nausea/Vomiting, mild, resolved without sequelae, unrelated, temporarily withdrawn
Feeling Hot (General disorders) | 0 (0) | 1 (1) — Feeling warm, moderate, resolved without sequelae, possible relatedness, permanently discontinued
Influenza like illness (General disorders) | 0 (0) | 1 (1) — Flu-like symptoms, moderate, ongoing at study exit, unrelated, no IP action taken
Fatigue (General disorders) | 2 (3) | 1 (1) — 4 total mild (4/4), resolved without sequelae (4/4), unrelated (1/4) unlikely (2/4), possible (1/4), no IP action taken (4/4)
Peripheral swelling (General disorders) | 1 (1) | 3 (3) — 4 total Swelling of legs/ankles (2/4) swelling of hands/feet (2/4), mild (4/4), resolved without sequelae (3/4) ongoing at study exit (1/4), unrelated (2/4) possible (2/4), no IP action taken (3/4) permanently discontinued (1/4)
Chest Pain (General disorders) | 1 (1) | 0 (0) — mild, resolved without sequelae, unrelated, no IP action taken
Asthenia (General disorders) | 1 (1) | 0 (0) — mild, resolved without sequelae, possible relatedness, temporarily withdrawn
Pain (General disorders) | 1 (1) | 0 (0) — Body aches, mild, resolved without sequelae, unrelated, temporarily withdrawn
Blood glucose increased (Investigations) | 1 (1) | 0 (0) — Elevated blood sugar, mild, ongoing at study exit, unlikely relatedness, no IP action taken
Heart rate irregular (Investigations) | 2 (2) | 2 (3) — 5 total irregular/fast heartbeat (5/5), mild (5/5), resolved without sequelae (4/5) ongoing at study exit (1/5), unrelated (2/5) unlikely (2/5) possible (1/5), no IP action taken (3/5) permanently discontinued (2/5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — mild, ongoing at study exit, unlikely relatedness, no IP action taken
Muscle cramps/spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — 2 total mild (1/2) severe (1/2), resolved without sequelae (2/2), unrelated (1/2) unlikely (1/2), no IP action taken (2/2)
Headache (Nervous system disorders) | 5 (6) | 2 (2) — 8 total mild (8/8), resolved without sequelae (7/8) ongoing at study exit (1/8), unrelated (4/8) unlikely (3/8) possible (1/8), no IP action taken (6/8) permanently discontinued (2/8)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) — 2 total mild (2/2), resolved without sequelae (2/2), possible relatedness (2/2), no IP action taken (2/2)
Vision blurred (Nervous system disorders) | 1 (1) | 0 (0) — Blurred vision/vision or hearing changes, mild, resolved without sequelae, unlikely relatedness, permanently discontinued
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) — cold/tingling/numb hands/feet, mild, resolved without sequelae, unrelated, no IP action taken
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) — 3 total mild (3/3), resolved without sequelae (1/3) resolved with sequelae (1/3) ongoing at study exit (1/3), unrelated (2/3) possible (1/3), no IP action taken (3/3)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cold symptoms, mild, ongoing at study exit, unrelated, no IP action taken
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) — 3 total mild (3/3), resolved without sequelae (1/3) resolved with sequelae (1/3) ongoing at study exit (1/3), unrelated (2/3) unlikely (1/3), no IP action taken (3/3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) — 6 total Breathing problems (6/6), mild (5/6) moderate (1/6), resolved without sequelae (3/6) resolved with sequelae (2/6) ongoing at study exit (1/6), unrelated (4/6) unlikely (2/6), no IP action taken (5/6) temporarily withdrawn (1/6)
Respiration Abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Breathing problem, severe, resolved without sequelae, unlikely relatedness, no IP action taken
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — 2 total Sweating (2/2), mild (2/2), resolved without sequelae (2/2), unrealted (2/2), no IP action taken (1/2) permanently discontinued (1/2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash, mild, resolved without sequelae, unlikely relatedness, no IP action taken
Dizziness (Vascular disorders) | 4 (4) | 1 (1) — 5 total Feeling faint/lightheadedness/falling (5/5), mild (4/5) moderate (1/5), resolved without sequelae (5/5), unlikely relatedness (2/5) possible (3/5), no IP action taken (5/5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT03640312/Prot_001.pdf
  • Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT03640312/SAP_002.pdf
  • Informed Consent Form (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT03640312/ICF_000.pdf